CLINICAL TRIAL: NCT00670800
Title: Influence of Insulin Resistance on Cognitive, Emotional and Opioid System Functioning in Women With Polycystic Ovary Syndrome
Brief Title: Study of Brain Function in Women With Insulin Resistant Polycystic Ovary Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Yolanda Smith, M.D., Professor, University of Michigan
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2276; HUM00008330 (Other: The University of Michigan IRBMED)
Record Dates: First submitted 2008-04-30; First posted 2008-05-02 (Estimated); Results first posted 2014-05-15 (Estimated); Last update posted 2014-05-21 (Estimated); Status verified 2014-05

CONDITIONS: Polycystic Ovary Syndrome
Keywords: Polycystic Ovary Syndrome; Insulin resistance; Metformin; Brain function
MeSH Terms: conditions — Polycystic Ovary Syndrome; Insulin Resistance | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Normal Controls (No Intervention): Control subjects will have 5 visits (screening, oral glucose tolerance test (OGTT), neuropsychological testing, functional magnetic resonance imaging (fMRI) and positron emission tomography (PET) as they will receive no treatment and will not have repeat studies. The baseline values obtained from the control subjects will be compared to the baseline values acquired from the PCOS affected subjects.
- PCOS Affected Women-Metformin Treatment (Experimental): Subjects with Polycystic Ovary Syndrome (PCOS) will be scheduled for 9 visits total: following the screening visit they will go through OGTT, neuro-psychological testing, fMRI and PET scan before and after 4 months of metformin use: 500mg tablets once daily with breakfast for 1 week, then increased to one tablet twice daily with breakfast & lunch for 1 week, then increased to one tablet three times daily with breakfast, lunch & dinner.
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Metformin — Following the baseline studies, PCOS affected women will be initiated on metformin at a dose of 500 mg orally after breakfast and the dose will be increased the following week to 500 mg twice daily (BID), adding a dose after lunch. On the third week, the dose will be increased to 500 mg three times daily (TID), adding a 500 mg tablet after supper. All subjects will be monitored for possible side effects such as nausea, vomiting, diarrhea, anorexia, and abdominal discomfort. These side effects tend to be mild, dose-related and improve with continued use of metformin. Hypoglycemia is rare and tends to occur in the setting of alcohol abuse or prolonged starvation. Malabsorption of vitamin B12 and folate occurs with long-term treatment, although it usually does not lead to anemia.
  Other Names: Glucophage
  Arms: PCOS Affected Women-Metformin Treatment

SUMMARY:
The purpose of this study is to evaluate the effects of insulin resistance on brain function in women with Polycystic Ovary Syndrome (PCOS). PCOS affected women will be evaluated prior to and following 4-month treatment with Metformin. Additionally, brain function in women with PCOS will be compared to the brain activity in normal control subjects with regular menstrual cycles.

DETAILED DESCRIPTION:
The pathogenesis of Polycystic Ovary Syndrome (PCOS), a reproductive and metabolic disorder, is associated with insulin resistance. The effects of insulin resistance on cognition, mood, opioid system and reproductive function in PCOS affected women are investigated in the current study. The identification of reversible changes in brain function and reproductive measures in insulin resistant PCOS patients would likely significantly influence treatment protocols for these young women.

1. Evaluate the differences in opioid tone in women with insulin resistant PCOS compared to normal controls.
2. Evaluate whether an oral hypoglycemic agent is capable of altering opioid tone in women with insulin resistant PCOS.

ELIGIBILITY:
Inclusion Criteria:

* Insulin-resistant PCOS (Arm: PCOS Affected Women)
* Irregular menstrual cycle (Arm: PCOS Affected Women)
* Hyperandrogenism (Arm: PCOS Affected Women)
* Regular menstrual cycles (Arm: Normal Controls)
* Normal hormonal levels (Arm: Normal Controls)
* Lack of hirsutism (Arm: Normal Controls)
* Acne-free (Arm: Normal Controls)
* Candidates are BMI-matched and screened for insulin resistance prior to inclusion. (Arm: Normal Controls)

Exclusion Criteria:

* Left handedness
* Acute medical illness
* Uncorrected thyroid disease
* Diabetes renal
* Cardiac or pulmonary insufficiency
* Active liver disease
* Neurological disease
* Current psychiatric illness
* Claustrophobia
* Contraindications to MRI
* Smoking
* Use of hormones
* Centrally acting or insulin sensitizing mediations
* Allergy to any opioid medication
* Substance abuse
* Pregnancy
* BMI >35.

Ages: 21 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2008-01; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yolanda R Smith, MD, MS, Principal Investigator — University of Michigan, Obstetrics and Gynecology
Locations (1):
- University of Michigan, Michigan Clinical Research Unit, Ann Arbor, Michigan, United States

REFERENCES:
- [Result] Berent-Spillson A, Love T, Pop-Busui R, Sowers M, Persad CC, Pennington KP, Eyvazaddeh AD, Padmanabhan V, Zubieta JK, Smith YR. Insulin resistance influences central opioid activity in polycystic ovary syndrome. Fertil Steril. 2011 Jun 30;95(8):2494-8. doi: 10.1016/j.fertnstert.2011.03.031. Epub 2011 Apr 12. PMID 21486668
- [Derived] Marsh CA, Berent-Spillson A, Love T, Persad CC, Pop-Busui R, Zubieta JK, Smith YR. Functional neuroimaging of emotional processing in women with polycystic ovary syndrome: a case-control pilot study. Fertil Steril. 2013 Jul;100(1):200-7.e1. doi: 10.1016/j.fertnstert.2013.02.054. Epub 2013 Apr 1. PMID 23557757

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Volunteers between the ages of 21 - 40 years were recruited from reproductive endocrinology clinic and newspapers. Women were excluded according to protocol exclusion criteria (see protocol)
Pre-assignment Details: Some potential subjects were excluded due to results of an oral glucose tolerance test (OGTT).
Groups:
- Women Affected With PCOS - Metformin: The Polycystic Ovary Syndrome (PCOS) affected group is comprised of subjects with insulin resistant PCOS, defined as having irregular menstrual cycles and hyperandrogenism with other causes ruled out. Insulin resistance will be identified as fasting homeostasis model assessment insulin resistance (HOMA2-IR) of 60%S or less.
- Women Controls Without PCOS: Control group is comprised of subjects without PCOS. These women have normal menstrual cycles and no evidence of insulin resistance (fasting HOMA2 IR of 80%S or more).
  .
  Exclusion criteria: left handedness, acute medical illness, uncorrected thyroid disease, diabetes, neurological disease, current psychiatric illness, smoking within the last 6 months, use of hormones within the last 2 months, pregnancy within the last 6 months, current or past history of substance abuse, use of corticosteroids (such as cortisol and prednisone), history of lactic acidosis (condition caused by the buildup of lactic acid in the body), heart, lung and kidney problems, liver disease, use of intravenous dyes, current cimetidine (Tagamet) use, use of medications that affect the brain (for example, codeine, anti-depressants, anti-psychotics).
Period: Overall Study
Arm/Group | Women Affected With PCOS - Metformin | Women Controls Without PCOS
Started | 7 | 7
Completed | 7 | 5 (Two controls were found to have insulin resistance and were excluded from analysis.)
Not Completed | 0 | 2
Not completed — 2 controls were insulin resistant | 0 | 2

BASELINE CHARACTERISTICS:
Population: Two controls were excluded from data analysis as they were later found to be insulin resistant.
Groups:
- PCOS Affected Women - Metformin: Right handed women who don't smoke and who drink very little will be considered eligible. Women with the following conditions (exclusion criteria) may not participate: left handedness, acute medical illness, uncorrected thyroid disease, diabetes, neurological disease, current psychiatric illness, smoking within the last 6 months, use of hormones within the last 2 months, pregnancy within the last 6 months, current or past history of substance abuse, use of corticosteroids (such as cortisol and prednisone), history of lactic acidosis (condition caused by the buildup of lactic acid in the body), heart, lung and kidney problems, liver disease, use of intravenous dyes, current cimetidine (Tagamet) use, use of medications that affect the brain (for example, codeine, anti-depressants, anti-psychotics).
- Normal Controls: Normal controls are matched for age and education and screened for insulin resistance. Controls will have HOMA2 IR of 80%S or greater, normal hormone levels, regular menstrual cycles, and lack hirsutism and acne. Exclusion criteria: Left handedness, acute medical illness, uncorrected thyroid disease, diabetes, neurological disease, current psychiatric illness, claustrophobia, contraindications to MRI (including pacemakers, pumps, surgical clips or metallic surgical devices), smoking within the last 6 months, use of hormones or insulin sensitizing mediation within the last 2 months, pregnancy within the last 6 months, current or past history of substance abuse, use of corticosteroids, cardiac or pulmonary insufficiency, active liver disease and transaminases elevations >2.5 X normal values, renal insufficiency (plasma creatinine level ≥1.4 mg/dl), use of centrally acting medications, allergy to any opioid medication, 300 lbs maximum weight limit (which is the max
- Total: Total of all reporting groups
Arm/Group | PCOS Affected Women - Metformin | Normal Controls | Total
Number analyzed (Participants) | 7 | 5 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 5 | 12
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.3 (4) | 26.6 (4) | 26.4 (4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 5 | 12
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 7 | 5 | 12
Weight [Median (Inter-Quartile Range); unit: pounds (lbs)] — Body weight measured in pounds (lbs)
  pounds (lbs) | 203.9 [161 to 246.8] | 123.7 [106 to 141.4] | 170.48 [138.1 to 202.9]
BMI (Body Mass Index) [Median (Inter-Quartile Range); unit: lbs/inch^2] — lbs/inches squared (pounds over inches squared)
  lbs/inch^2 | 35.3 [19.1 to 51.5] | 23 [19.9 to 26.1] | 29.5 [22.95 to 37.75]
Waist Circumference [Median (Inter-Quartile Range); unit: cm] — Waist circumference measured in cm
  cm | 102 [74.4 to 129.6] | 72 [58.5 to 85.5] | 92 [73.5 to 103.5]
Free Testosterone [Median (Inter-Quartile Range); unit: pg/ml] — Free testosterone measured in picograms over milliliters
  pg/ml | 1.5 [0.6 to 2.4] | .5 [0.3 to 0.7] | 1 [0.525 to 1.4]
Total Testosterone [Median (Inter-Quartile Range); unit: ng/ml] — Total Testosterone measured in nanograms over milliliters
  ng/ml | .7 [.19 to 1.21] | .36 [.04 to .68] | .55 [.37 to .825]
Total Cholesterol [Median (Inter-Quartile Range); unit: mg/dl] — Total cholesterol measured in milligrams over deciliter
  mg/dl | 157 [111 to 203] | 179 [119 to 239] | 174 [140.25 to 195]
DHEAS [Median (Inter-Quartile Range); unit: ug/dl] — Dehydroepiandrosterone Sulfate (DHEAS)measured in micrograms/deciliter
  ug/dl | 200 [112 to 288] | 189 [101 to 277] | 191 [145 to 236.5]
HDL [Median (Inter-Quartile Range); unit: mg/dl] — High-density lipoprotein measured in milligrams/deciliter
  mg/dl | 47 [30 to 64] | 76 [52 to 100] | 55.5 [47 to 76]
Triglycerides [Median (Inter-Quartile Range); unit: mg/dl] — Triglycerides measured in measured in milligrams/deciliter
  mg/dl | 74 [32 to 116] | 72 [45 to 109] | 73 [59.75 to 112.25]
Fasting Insulin [Median (Inter-Quartile Range); unit: uU/ml] — Fasting Insulin measured in microunits/milliliter
  uU/ml | 21.4 [16.3 to 26.5] | 8.1 [7.2 to 9] | 17.25 [8.475 to 21.475]
Fasting Glucose [Median (Inter-Quartile Range); unit: mg/dl] — Fasting Glucose measured in milligrams/deciliter
  mg/dl | 87 [72 to 102] | 89 [82 to 96] | 89 [85.25 to 95.75]
Homeostatic Model Assessment (HOMA) [Median (Inter-Quartile Range); unit: % - percentage] — Homeostatic model assessment sensitivity reported in percentage
  % - percentage | 36.6 [27.3 to 45.9] | 95.4 [82.6 to 108.2] | 46.65 [36.375 to 91.025]
HOMA-IR [Median (Inter-Quartile Range); unit: mU/L] — Homeostatic model assessment insulin resistance measured in milliunits per Liters
  mU/L | 2.7 [2.1 to 3.3] | 1 [.8 to 1.2] | 2.150 [1.1 to 2.775]

OUTCOME MEASURES:

1. Primary Outcome: Mu-opioid Binding Potential Measured in Left Nucleus Accumbens
Description: Mu-opioid binding potential in left nucleus accumbens is measured before and after 4 months of Metformin treatment.
  Mu-opioid binding potential is measured in vivo with C11-carfentanil positron emission tomography in women with PCOS before and after 4 months of metformin treatment.
  Binding Potential is measured by the ratio of Mu-opioid receptor concentration (Bmax)/Receptor radiotracer (C11-carfentanil) affinity (Kd.)
  Control group was measured at baseline only.
Time Frame: Baseline and after 4 months
Population: All 7 PCOS women completed the protocol and were included. 5 of 7 controls were included in this analysis. 2 controls were excluded from analysis because repeat baseline OGTT showed HOMA %S of <80%.
Measure: Mean (Standard Deviation); unit: ratio
Groups:
- PCOS Affected Women Pre-Metformin (Baseline); PCOS Affected Women Post-Metformin (After 4 Months): PCOS will be defined as meeting the criteria of irregular menstrual cycles and hyperandrogenism (on physical exam or laboratory testing), with other causes ruled out. Subjects with insulin resistant PCOS must meet criteria for insulin resistance based on the 2 hr OGTT (Oral Glucose Tolerance Test). Insulin resistance will be defined as fasting HOMA2 IR of 60%S or less.
- Normal Controls: Normal controls will have HOMA2 IR of 80%S or greater, normal hormone levels, regular menstrual cycles (range 24 - 34 days), and lack hirsutism and acne. Control subjects are matched for age and education with the PCOS affected women. Control data is measured once (at baseline time frame) for the entire study.
Arm/Group | PCOS Affected Women Pre-Metformin (Baseline) | PCOS Affected Women Post-Metformin (After 4 Months) | Normal Controls
Number analyzed (Participants) | 7 | 7 | 5
ratio | 1.95 (0.17) | 1.65 (.27) | 1.53 (0.28)
Statistical Analysis 1: Comparison: PCOS Affected Women Pre-Metformin (Baseline) vs Normal Controls; Test type: Superiority or Other; p = 0.143, t-test, 2 sided
Statistical Analysis 2: Comparison: PCOS Affected Women Post-Metformin (After 4 Months) vs Normal Controls; Test type: Superiority or Other; p = 0.900, t-test, 2 sided
Statistical Analysis 3: Comparison: PCOS Affected Women Pre-Metformin (Baseline) vs PCOS Affected Women Post-Metformin (After 4 Months); Test type: Superiority or Other; p = 0.133, t-test, 2 sided

2. Primary Outcome: Mu-opioid Binding Potential Measured in Right Nucleus Accumbens
Description: Mu-opioid binding potential in right nucleus accumbens measured before and after 4 months of Metformin treatment.
  Mu-opioid binding potential is measured in vivo with C11-carfentanil positron emission tomography in women with PCOS before and after 4 months of metformin treatment.
  Binding Potential is measured by the ratio of Mu-opioid receptor concentration (Bmax)/Receptor radiotracer (C11-carfentanil) affinity (Kd.)
  Control group was measured at baseline only.
Time Frame: Baseline and after 4 months
Population: All 7 PCOS women were included, 2 controls were excluded because repeat baseline HOMA2-IR %S was <80%.
Measure: Mean (Standard Deviation); unit: ratio
Groups:
- Normal Control Women: Normal controls will have HOMA2 IR of 80%S or greater, normal hormone levels, regular menstrual cycles (range 24 - 34 days), and lack hirsutism and acne. Control subjects are matched for age and education with the PCOS affected women. Control data is measured once (at baseline time frame) for the entire study.
Arm/Group | PCOS Affected Women Pre-Metformin (Baseline) | PCOS Affected Women Post-Metformin (After 4 Months) | Normal Control Women
Number analyzed (Participants) | 7 | 7 | 5
ratio | 2.40 (.11) | 2.11 (0.21) | 2.05 (0.28)
Statistical Analysis 1: Comparison: PCOS Affected Women Pre-Metformin (Baseline) vs Normal Control Women; Test type: Superiority or Other; p = 0.049, t-test, 2 sided
Statistical Analysis 2: Comparison: PCOS Affected Women Post-Metformin (After 4 Months) vs Normal Control Women; Test type: Superiority or Other; p = 0.717, t-test, 2 sided
Statistical Analysis 3: Comparison: PCOS Affected Women Pre-Metformin (Baseline) vs PCOS Affected Women Post-Metformin (After 4 Months); Test type: Superiority or Other; p = 0.038, t-test, 2 sided

3. Primary Outcome: Mu-opioid Binding Potential Measured in Left Amygdala
Description: Mu-opioid binding potential in left amygdala measured before and after 4 months of Metformin treatment.
  Mu-opioid binding potential is measured in vivo with C11-carfentanil positron emission tomography in women with PCOS before and after 4 months of metformin treatment.
  Binding Potential is measured by the ratio of Mu-opioid receptor concentration (Bmax)/Receptor radiotracer (C11-carfentanil) affinity (Kd.)
Time Frame: Baseline and after 4 months
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | PCOS Affected Women Pre-Metformin (Baseline) | PCOS Affected Women Post-Metformin (After 4 Months) | Normal Controls
Number analyzed (Participants) | 7 | 7 | 5
ratio | 2.28 (.17) | 2.08 (.19) | 2.03 (.07)
Statistical Analysis 1: Comparison: PCOS Affected Women Pre-Metformin (Baseline) vs Normal Controls; Test type: Superiority or Other; p = 0.498, t-test, 2 sided
Statistical Analysis 2: Comparison: PCOS Affected Women Post-Metformin (After 4 Months) vs Normal Controls; Test type: Superiority or Other; p = 0.835, t-test, 2 sided
Statistical Analysis 3: Comparison: PCOS Affected Women Pre-Metformin (Baseline) vs PCOS Affected Women Post-Metformin (After 4 Months); Test type: Superiority or Other; p = 0.606, t-test, 2 sided

4. Primary Outcome: Mu-opioid Binding Potential Measured in Right Amygdala
Description: Mu-opioid binding potential in right amygdala measured before and after 4 months of Metformin treatment.
  Mu-opioid binding potential is measured in vivo with C11-carfentanil positron emission tomography in women with PCOS before and after 4 months of metformin treatment.
  Binding Potential is measured by the ratio of Mu-opioid receptor concentration (Bmax)/Receptor radiotracer (C11-carfentanil) affinity (Kd.)
  Control group was measured at baseline only.
Time Frame: Baseline and 4 months
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | PCOS Affected Women Pre-Metformin (Baseline) | PCOS Affected Women Post-Metformin (After 4 Months) | Normal Controls
Number analyzed (Participants) | 7 | 7 | 5
ratio | 2.28 (.23) | 2.11 (.22) | 2.06 (.26)
Statistical Analysis 1: Comparison: PCOS Affected Women Pre-Metformin (Baseline) vs Normal Controls; Test type: Superiority or Other; p = 0.118, t-test, 2 sided
Statistical Analysis 2: Comparison: PCOS Affected Women Post-Metformin (After 4 Months) vs Normal Controls; Test type: Superiority or Other; p = 0.581, t-test, 2 sided
Statistical Analysis 3: Comparison: PCOS Affected Women Pre-Metformin (Baseline) vs PCOS Affected Women Post-Metformin (After 4 Months); Test type: Superiority or Other; p = 0.190, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Adverse events were followed in the course of 2 years.
Groups:
- Normal Controls: Women without PCOS
- PCOS Affected Women on Metformin: Women with PCOS and insulin resistance
Arm/Group | Normal Controls | PCOS Affected Women on Metformin
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/7
Other Adverse Events (participants affected / at risk) | 1/5 | 1/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Normal Controls (N=5) | PCOS Affected Women on Metformin (N=7)
High Glucose During Oral Glucose Tolerance Test (OGTT) (Metabolism and nutrition disorders) | 0 (0) | 1 (1) — OGTT after 3 ½ months of Metformin. This event was unexpected as Metformin is prescribed to reduce the blood sugar levels and is a widely accepted anti-diabetic drug.
Nausea from Carfentanil at PET (General disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No